CLINICAL TRIAL: NCT04458610
Title: BTK Inhibitor Zanubrutinib (BGB-3111) in Combination With Rituximab for Previously Untreated Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Zanubrutinib and Rituximab for the Treatment of Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0012; NCI-2020-05053 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0012 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; CT-P10; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (zanubrutinib, rituximab) (Experimental): See Detailed Description.
  Interventions: Biological: Rituximab; Drug: Zanubrutinib

INTERVENTIONS:
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Zanubrutinib — Given PO
  Other Names: BGB-3111; Brukinsa; BTK-InhB

SUMMARY:
This phase II trial studies how well zanubrutinib and rituximab work in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma for which the patient has not received treatment in the past (previously untreated). Zanubrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. The study is being done to find out if zanubrutinib combined with rituximab can help control previously untreated chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of patients who have treatment-free remission 6 months after discontinuation of zanubrutinib.

SECONDARY OBJECTIVES:

I. To determine clinical factors associated with a treatment-free remission of more than 6 months after discontinuation of zanubrutinib.

II. To determine the treatment-free remission length. III. To evaluate the efficacy of re-treatment with zanubrutinib plus rituximab in patients who relapse.

OUTLINE:

FRONTLINE THERAPY: Patients receive zanubrutinib orally (PO) twice daily (BID) on days 1-28. Patients also receive rituximab intravenously (IV) over 3-4 hours on days 1, 8, 15, and 22 of cycle 1 and on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 7, patients with complete response (CR) continue zanubrutinib PO BID on days 1-28 for up to 6 additional cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 7, patients with partial response (PR) or stable disease (SD) continue zanubrutinib PO BID on days 1-28 and rituximab IV over 3-4 hours on day 1 for up to 6 additional cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 13, patients with CR continue zanubrutinib PO BID on days 1-28 for up to 6 additional cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 13, patients with PR or SD continue zanubrutinib PO BID on days 1-28 for up to 12 additional cycles in the absence of disease progression or unacceptable toxicity. Patients who do not have a PR after 24 cycles either continue zanubrutinib if there is a clinical benefit, or pursue alternative therapy per treating physician discretion.

RE-TREATMENT FOR RELAPSED DISEASE: Patients with disease relapse and active disease that requires salvage therapy may restart zanubrutinib PO BID on days 1-28 and rituximab IV over 3-4 hours on day 1. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 7, patients continue zanubrutinib PO BID on days 1-28 for up to 18 additional cycles in the absence of disease progression or unacceptable toxicity and then discontinue if in CR. Beginning cycle 25, patients with PR or SD may continue zanubrutinib PO BID on days 1-28 for up to 36 additional cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 60 days, and then every 120 days for up to 5 years or until disease progression or start of a new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) and be previously untreated
* Patients must have an indication for treatment by 2018 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria
* Patients must understand and voluntarily sign an informed consent, and be able to comply with study procedures and follow-up examinations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients of childbearing potential must be willing to practice highly effective birth control (e.g., condoms, implants, injectables, combined oral contraceptives, intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the study and for 30 days after the last dose of study drug. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) except for patients with bilirubin elevation due to Gilbert's disease who will be allowed to participate
* An alanine aminotransferase (ALT) =< 2.5 x ULN
* An estimated creatinine clearance (CrCl) of > 30 mL/min, as calculated by the Cockcroft-Gault equation unless disease related
* Free of prior malignancies for 3 years with exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. If patients have another malignancy that was treated within the last 3 years, such patients can be enrolled, after consultation with the principal investigator, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy
* A urine pregnancy test (within 7 days of day 1) is required for women with childbearing potential

Exclusion Criteria:

* Pregnant or breast-feeding females
* Prior therapy with zanubrutinib or other kinase inhibitors that target BCR signaling (such as ibrutinib, idelalisib)
* Prior CLL-directed treatment including chemotherapy, chemo-immunotherapy, monoclonal antibody therapy, radiotherapy, high-dose corticosteroid therapy (more than 60 mg prednisone daily or equivalent), or immunotherapy within 21 days prior to enrollment or concurrent with this trial. Patients that receive zanubrutinib salvage therapy cannot have received any other CLL-directed therapy besides frontline zanubrutinib plus rituximab
* Investigational agent received within 30 days prior to the first dose of study drug. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to grade 1 or less prior to first dose of study drug
* Systemic fungal, bacterial, viral, or other infection not controlled by antimicrobial therapy, in the assessment of the treating physician(s) and/or the principal investigator
* Patients with uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP), i.e. with laboratory signs of active hemolysis or thrombocytopenia, requiring support with blood products and/or with rapid decline in hemoglobin (> 1 gram/dL per day) or platelet counts (> 10,000/uL per day)
* Patients with severe hematopoietic insufficiency, as defined by an absolute neutrophil count of less than 500/uL, unless disease-related, and/or a platelet count of less than 30,000/uL at time of screening for this protocol
* Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo therapy with zanubrutinib and rituximab
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Patients with a history of paroxysmal atrial fibrillation (PAF) or deep vein thrombosis or pulmonary embolism (DVT/PE) can be included if they had no signs of PAF or DVT/PE in the last 6 months before enrolment. Patients with ongoing atrial fibrillation (AFib) or ongoing PAF or DVT/PE should be excluded
* History of stroke or cerebral hemorrhage within 6 months
* Evidence of bleeding diathesis or coagulopathy within 3 months
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 1. Bone marrow aspiration and/or biopsy are allowed
* Serious, non-healing wound, ulcer, or bone fracture
* Treatment with warfarin (Coumadin) or any other vitamin K antagonist. Patients who recently received warfarin must be off warfarin for at least 7 days prior to start of the study. Patients receiving novel oral anticoagulant (NOAC), also termed direct oral anticoagulant (DOAC) are permitted to enroll. Patients who are currently on a vitamin K antagonist must be switched to a non-vitamin K antagonist, such as a NOAC/DOAC
* Patients with active hepatitis B (hepatitis B virus [HBV]) or hepatitis C
* Patients with known human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Success rate | At 6 months after discontinuation of zanubrutinib
  Will estimate the proportion of patients who have treatment-free remission 6 months after discontinuation of zanubrutinib. Success rate will be estimated with 95% credible interval and confidence interval.

SECONDARY OUTCOMES:
Clinical factors associated with a treatment-free remission of more than 6 months after discontinuation of zanubrutinib | Up to 5 years after discontinuation of zanubrutinib
  To assess the contribution of various factors to relapse risk, will use Cox's proportional hazards analysis of predictors that have a p value < 0.2 in the univariate analysis.
Treatment-free remission length | Up to 5 years after discontinuation of zanubrutinib
  The median treatment-free remission duration will be calculated by Kaplan-Meier analysis, and stratified groups will be compared with the log-rank test.
Overall response | After 6 cycles of treatment (each cycle is 28 days)
  Defined as complete response or partial response after patients received 6 cycles of treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Burger, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org